CLINICAL TRIAL: NCT06873490
Title: Evaluation of the External Apical Root Resorption and the Periodontal Indices After the En-masse Retraction of the Upper Anterior Teeth Stimulated by Low-intensity Electrical Stimulation: a Randomized Controlled Trial
Brief Title: External Root Resorption and Periodontal Status During Retraction of the Upper Anterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-2-2025
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric stimulation with retraction (Experimental): Electric current will be applied in this group of patients using a removable device.
  Interventions: Device: Electric stimulation removabel device
- Traditional retraction (Active Comparator): No acceleration method will be performed in this group. Only the traditional method of retraction will be followed.
  Interventions: Procedure: Traditional retraction method.

INTERVENTIONS:
Device: Electric stimulation removabel device — The device will be used to stimulate orthodontic tooth movement through a specific design used to deliver the current to the mucosa around the teeth being retracted.
  Arms: Electric stimulation with retraction
Procedure: Traditional retraction method. — In this intervention, the upper anterior teeth will be retracted together backward using the traditional retraction method. No acceleration devices will be used in conjunction with this procedure.
  Arms: Traditional retraction

SUMMARY:
This RCT will include 34 patients requiring en-masse retraction of upper anterior teeth after maxillary first premolars extraction.

Patients accepted into the study will be randomly assigned to one of two groups in a 1:1 allocation ratio: the electrically stimulated en-masse retraction group (ESER) and the conventional en-masse retraction group (CER). In both groups, the upper anterior teeth will be retracted en masse by applying 250 g of force on each side using closed nickel-titanium coil springs. Mini-implants will be used to provide the maximum anchorage.

The outcomes of the study will be the external apical root resorption (EARR) and the periodontal status of the upper anterior teeth during the treatment stages.

DETAILED DESCRIPTION:
Young adult patients who visit the Department of Orthodontics at Damascus University-Faculty of Dentistry during the sample collection period will be examined to determine the orthodontic treatment plan. Written informed consent will be obtained from all patients who meet the inclusion criteria and accept to participate in the trial.

Before starting the leveling and alignment procedures on the maxillary dental arch, skeletal anchorage will be secure on the maxillary dental arch using self-drilling mini-implants (1.6 * 8 mm; 3S screw, Hubit™, Seoul, Korea) that will apply between the roots of the maxillary first molars and the second premolars. The patients will be referred for maxillary first premolars extraction at the Department of Maxillofacial Surgery, Damascus University, Faculty of Dentistry.

This study will use fixed orthodontic appliances with an MBT prescription and a 0.022-inch bracket slot (VotionTM, Ortho Technology, Florida, USA). The two groups will follow a uniform wire sequence starting from a 0.014-inch NiTi wire until they reach the 0.019*0.025-inch stainless steel basic archwire, with a 3-week interval between each wire.

The sliding technique will be used for en-masse retraction in both study groups. An orthodontic force of approximately 500 g (250 g on each side) will be applied to the crimpable hooks using bilateral closed coil nickel titanium springs (NT3 closed coil springs, American Orthodontics, Sheboygan, Wisconsin) anchored to orthodontic mini-screws. Patients will be followed up every 2 weeks during this phase to adjust the springs to maintain a constant force. The endpoint of en-masse retraction in both groups will be determined when the maxillary canines achieve a Class I relationship with the mandible and a normal incisor relationship.

The removable electrical stimulation device utilized in the study by Shaadouh et al.. to provide the electrical stimulation will be used in this trial for the same purpose.

Each patient in the low-intensity electrical stimulation group will be asked to wear a removable device for five hours daily until the completion of the retraction of the upper anterior teeth.

To evaluate external apical root resorption (EARR), digital panoramic radiographs will be taken at three time points: before orthodontic treatment (T0), before en-masse retraction (T1), and after en-masse retraction (T2). The ImageJ software (NIH and LOCI, Madison, Wisconsin, USA) was used to analyze these radiographs. The method, originally described by Linge and Linge will be used to calculate the root resorption.

The gingival index (GI), the papillary bleeding index (PBI), and the dental plaque index (DPI) will be measured on the upper anterior teeth at the previous assessment times.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult patients, Male and female, Age range: 18-25 years.
2. Class II Division 1 malocclusion :

   * Mild/moderate skeletal Class II (ANB= 5-7 degrees)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
3. Permanent occlusion.
4. The Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement, such as corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs).
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   Probing depth ≥ 4 mm Radiographic evidence of bone loss Gingival index > 1 Plaque index > 1
5. Patient had previous orthodontic treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Change in external apical root resorption | The digital panoramic radiographs will be taken at: (T1) one day before treatment commencement, (T2) at the end of the levelling stage (expected to occur within 3 - 4 months), (T3) one day after the end of retraction (expected to occur within 6 months).
  The root length will be measured for each root of six upper anterior teeth. The method originally described by Linge and Linge will be used. The amount of root resorption (in millimeters) will be calculated using the following equation: Root Resorption = Root Length (T0) - (Root Length (T1) × Correction Factor). The Correction Factor will be calculated by dividing the crown Length (T0) to the crown Length (T1).

SECONDARY OUTCOMES:
Change in the Gingival Index | Evaluation will be performed at: (T1) one day before treatment commencement, (T2) at the end of the levelling stage (expected to occur within 3 - 4 months), (T3) one day after the end of retraction (expected to occur within 6 months).
  Assessment will be performed using a gingival probe according to Silness and Loe.
  (0) = Normal gingiva.
  1. = Mild inflammation: slight color change, slight edema. No bleeding on probing.
  2. = Moderate inflammation: redness, edema and glazing. Bleeding on probing.
  3. = Sever inflammation: marked redness and edema, ulceration, and tendency to spontaneous bleeding
Change in the Dental Plaque index | Evaluation will be performed at: (T1) one day before treatment commencement, (T2) at the end of the levelling stage (expected to occur within 3 - 4 months), (T3) one day after the end of retraction (expected to occur within 6 months).
  Assessment will be performed using a gingival probe according to Silness and Loe.
  (0) = No plaque.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after disclosing solution or using the probe on the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin, which can be seen with the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or the tooth and gingival margin.
Change in the Bleeding Index | Evaluation will be performed at: (T1) one day before treatment commencement, (T2) at the end of the levelling stage (expected to occur within 3 - 4 months), (T3) one day after the end of retraction (expected to occur within 6 months).
  The Bleeding index will be used to assess the status of periodontal tissues and the amount of congestion in the gingival margins around the anterior teeth.
  According to Muhlemann, an assessment will be performed using a gingival probe. (0) = No bleeding.
  1. = A single discrete bleeding point appears.
  2. = Several isolated bleeding points or a single fine line of blood appears.
  3. = The interdental triangle fills with blood shortly after probing.
  4. = Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
Change in Gingival Recession | Evaluation will be performed at: (T1) one day before treatment commencement, (T2) at the end of the levelling stage (expected to occur within 3 - 4 months), (T3) one day after the end of retraction (expected to occur within 6 months).
  This will be measured in millimeters from the cement-enamel junction to the gingival margin level around the six anterior teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Rashad Ibrahem Shaadouh, DDS MSc, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaadouh RI, Hajeer MY, Al-Sabbagh R, Alam MK, Mahmoud G, Idris G. A Novel Method to Accelerate Orthodontic Tooth Movement Using Low-Intensity Direct Electrical Current in Patients Requiring en-Masse Retraction of the Upper Anterior Teeth: A Preliminary Clinical Report. Cureus. 2023 May 24;15(5):e39438. doi: 10.7759/cureus.39438. eCollection 2023 May. PMID 37234453
- [Background] Davidovitch Z, Finkelson MD, Steigman S, Shanfeld JL, Montgomery PC, Korostoff E. Electric currents, bone remodeling, and orthodontic tooth movement. II. Increase in rate of tooth movement and periodontal cyclic nucleotide levels by combined force and electric current. Am J Orthod. 1980 Jan;77(1):33-47. doi: 10.1016/0002-9416(80)90222-5. PMID 6243448
- [Background] Spadari GS, Zaniboni E, Vedovello SA, Santamaria MP, do Amaral ME, Dos Santos GM, Esquisatto MA, Mendonca FA, Santamaria M Jr. Electrical stimulation enhances tissue reorganization during orthodontic tooth movement in rats. Clin Oral Investig. 2017 Jan;21(1):111-120. doi: 10.1007/s00784-016-1759-6. Epub 2016 Feb 26. PMID 26917494
- [Background] Shaadouh RI, Hajeer MY, Awawdeh MA, Jaber ST, Mahmoud GA, Almasri IA. Effectiveness of low-intensity electrical current in accelerating the en-masse retraction of the upper anterior teeth following first-premolar extraction in young adult patients with Class II division 1 malocclusion: A randomized controlled clinical trial. Int Orthod. 2024 Dec;22(4):100921. doi: 10.1016/j.ortho.2024.100921. Epub 2024 Sep 23. PMID 39316889
- [Derived] Shaadouh RI, Hajeer MY, Alam MK, Jaber ST. Effect of Low-Intensity Electrical Stimulation on External Apical Root Resorption and Periodontal Indices Following En-Masse Retraction of Upper Anterior Teeth in Young Adults: A Randomized Controlled Trial. Clin Exp Dent Res. 2025 Aug;11(4):e70188. doi: 10.1002/cre2.70188. PMID 40762524